CLINICAL TRIAL: NCT01417234
Title: Post-Market Clinical Evaluation of the Spiracur SNaP Wound Care System for Treatment of Acute Trauma and Acute Surgical Excision Wounds
Status: Completed | Type: Observational
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: 102110
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Trauma-related Wound; Surgical Wound, Recent
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SNaP® Wound Care System
  Interventions: Device: SNaP® Wound Care System

INTERVENTIONS:
Device: SNaP® Wound Care System — Wound dressing applications using customized system. Dressing applications changes per manufacturer recommendation.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Spiracur SNaP® Wound Care System for the treatment of acute trauma and acute surgical excision wounds. The secondary purpose will be to compare the prospective patients to retrospectively treated acute trauma wounds to further evaluate efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Trauma wound, pressure ulcer, post operative wound, colostomy take-down site, or other acute wound deemed appropriate by study investigator(s) as the source of the wound on any part of the body including head and neck, torso, and extremities
* Wound < 16 cm in greatest diameter
* Subject ≥ 18 years of age
* Exudate < 25 ml/ day (estimate)
* Female subjects of child-bearing potential must be willing to take a urine pregnancy test prior to starting study
* Subject is willing and able to sign informed consent

Exclusion Criteria:

* Wound > 45 days old
* Wound-related cellulitis
* Wound located in an area not amenable to forming an air-tight seal
* Subject has untreated osteomyelitis
* Subject is allergic to wound care products
* Wound has exposed blood vessels not suitable for negative pressure therapy
* Subject is pregnant
* Subject is actively participating in other clinical trials that conflict with current study
* Subject has fistulas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from exisiting investigator patient population.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNaP® Wound Care System
Started | 30
Completed | 27
Not Completed | 3
Not completed — Subject non-compliant | 3

BASELINE CHARACTERISTICS:
Arm/Group | SNaP® Wound Care System
Number analyzed (Participants) | 30
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 55 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12
  Unknown | 18
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Wound Closure
Description: Percent of subjects with study wound deemed closed at 12 weeks
  1 wound is studied per participant
Time Frame: 12 weeks
Population: Per protocol population used for analysis. 3 subjects withdrew from study early due to non-compliance with study therapy and were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | SNaP® Wound Care System
Number analyzed (Participants) | 27
Participants | 22

2. Secondary Outcome: Percent Wound Size Change
Description: Percent change in wound size from baseline to week 4 (Week 4 - baseline / baseline)
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SNaP® Wound Care System
Number analyzed (Participants) | 30
percent change | -41 (0.43)

3. Secondary Outcome: Percent Wound Size Change
Description: Percent change in wound size from week 4 to week 8 (Week 8 - Week 4 / Week 4)
Time Frame: 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SNaP® Wound Care System
Number analyzed (Participants) | 30
percent change | -18.2 (0.39)

4. Secondary Outcome: Percent Wound Size Change
Description: Percent change in wound size from week 8 to week 12 (12 Weeks - 8 weeks / 8 weeks)
Time Frame: 8 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SNaP® Wound Care System
Number analyzed (Participants) | 30
percent change | -3.6 (0.11)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | SNaP® Wound Care System
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No